CLINICAL TRIAL: NCT06838559
Title: Multicentre, Randomized, Controlled Clinical Trial on 7-day Followed by Maintenance Therapy for 10 Weeks vs. 14-day and no Maintenance Course of Prednisolone for the Treatment of Infantile Epileptic Spasms Syndrome (IESS)
Brief Title: Clinical Trial on 7-day Followed by Maintenance Therapy for 10 Weeks vs. 14-day and no Maintenance Course of Prednisolone for the Treatment of Infantile Epileptic Spasms Syndrome (IESS)
Acronym: SLISS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colombo (Other)
Responsible Party: Principal Investigator, Jithangi Wanigasinghe, Professor in Paediatric Neurology, Department of Paediatrics, Faculty of Medicine, University of Colombo, Sri Lanka, University of Colombo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-24-125; U1111-1318-1599 (Other: WHO ICTRP)
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Spasms, Infantile; Prednisolone
Keywords: Randomized controlled trial; Spasms, Infantile; Prednisolone; Infant; Electroencephalography; Child Development; Relapse; Tapering Regimen; Treatment Duration
MeSH Terms: conditions — Spasms, Infantile; Recurrence

STUDY DESIGN:
Intervention Model Description: Randomized (1:1), single-blinded, multi-centre, parallel-group clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Both the outcome assessor (MBBS-qualified research assistant) and the data analyst will be blinded to the treatment arms. By implementing these measures, the risk of bias is minimized, and the credibility of the study results is enhanced, ensuring that the conclusions drawn from the data are based solely on the observed effects of the treatments without any influence from knowledge of the treatment allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment arm A (Experimental): The initial phase of the intervention involves administering prednisolone orally at a dosage of 10 mg, four times daily (40 mg/day) for 7 days. This will be followed by a tapering regimen over 15 days (~2 weeks) as outlined below:
  10 mg three times daily - 5 days 10 mg twice daily - 5 days 10 mg daily - 5 days The second phase of the intervention begins at the end of 15 days, where a prolonged tapering of prednisolone at a low dose (<0.4 mg/kg per day) will be administered as 10 mg once daily, twice a week, for an additional 10 weeks.
  Interventions: Drug: Short-Duration Oral Prednisolone with Extended Tapering
- treatment arm B (Active Comparator): Prednisone will be administered orally at a dose of 10 mg, four times daily (40 mg/day) for 14 days. This is the standard therapy currently given to children with IESS in Sri Lanka. This will be followed by a tapering regimen over 15 days (~2 weeks) as outlined below:
  10 mg three times daily - 5 days 10 mg twice daily - 5 days 10 mg daily - 5 days No additional tapering will be implemented.
  Interventions: Drug: Standard Oral Prednisolone Regimen with Tapering

INTERVENTIONS:
Drug: Short-Duration Oral Prednisolone with Extended Tapering — In treatment arm A, oral prednisolone will be administered in tablet form (5 mg strength) as follows: an initial phase of 10 mg four times daily (total 40 mg/day) for 7 days, followed by a 15-day tapering phase-10 mg three times daily for 5 days, 10 mg twice daily for 5 days, and 10 mg once daily for 5 days. After tapering, a prolonged low-dose maintenance phase will be implemented, where 10 mg is given once daily twice a week for an additional 10 weeks. This regimen is designed to test whether a shorter high-dose course, combined with extended low-dose maintenance, can provide equivalent control of infantile epileptic spasms syndrome while reducing the adverse effects associated with longer high-dose therapy, compared to the standard 14-day high-dose regimen (treatment arm B).
  Arms: treatment arm A
Drug: Standard Oral Prednisolone Regimen with Tapering — Prednisone oral tablets, 10 mg, administered four times daily (40 mg/day) for 14 days, followed by a tapering phase over 15 days: 10 mg three times daily for 5 days, 10 mg twice daily for 5 days, and 10 mg once daily for 5 days. No further tapering will be implemented after the initial 14-day treatment period. This regimen represents the standard therapy for Infantile Spasms in Sri Lanka.
  Arms: treatment arm B

SUMMARY:
The goal of this clinical trial is to learn if short courses (7 days) of oral prednisolone are as effective as longer courses (14 days) in treating Infantile Epileptic Spasms Syndrome (IESS) in infants. The main questions it aims to answer are:

1. Does a 7-day course of oral prednisolone result in a similar or better reduction in spasm frequency compared to a 14-day course?
2. Does the duration of treatment (7 vs. 14 days) influence relapse rates and developmental outcomes in infants with IESS?
3. Researchers will compare the effects of the two treatment arms (7-day course vs. 14-day course of oral prednisolone) to see if there is a difference in efficacy and safety.

Participants will:

1. Receive either a 7-day or 14-day course of oral prednisolone as part of their treatment
2. Be monitored for spasm frequency and any side effects during hospital observation for the first 48 hours
3. Maintain a spasm diary during the treatment period to track spasm frequency
4. Return for follow-up visits at 7 days, 14 days, 28 days, 42 days, 3 months, 6 months, and 12 months to assess treatment response, relapse, and developmental outcomes

DETAILED DESCRIPTION:
Study Title: Comparison of Short (7-Day) versus Long (14-Day) Courses of Oral Prednisolone in the Treatment of Infantile Epileptic Spasms Syndrome (IESS)

Study Overview: This is a clinical trial designed to compare the efficacy and safety of two treatment regimens using oral prednisolone for infants with Infantile Epileptic Spasms Syndrome (IESS). The study aims to evaluate the impact of treatment duration (7 days vs. 14 days) on spasm resolution, relapse rates, and developmental outcomes in infants with IESS. Participants will be randomized into two treatment arms to receive either a 7-day or 14-day course of oral prednisolone, and they will be followed for a year to assess outcomes related to spasm control, relapse, adverse effects, and long-term development.

Study Population: The study will include infants diagnosed with IESS, aged 3 to 24 months, who are receiving care at participating clinical sites. Eligibility criteria ensure the inclusion of infants with confirmed spasms, with or without known aetiology, and those who have not previously received systemic treatment for IESS.

Objectives:

* Primary Objective: To compare the effectiveness of 7-day versus 14-day oral prednisolone treatment in reducing spasm frequency in infants with IESS.
* Secondary Objectives: To evaluate the impact of treatment duration on relapse rates, developmental outcomes, and adverse effects.
* Exploratory Objectives: To assess any differences in long-term neurodevelopmental progress, including cognitive and motor development, and to compare EEG findings between treatment groups.

Methodology:

1. Randomization: Participants will be randomly assigned to receive either 7 days or 14 days of oral prednisolone, with blinding for the treatment duration.
2. Treatment Regimen:

   * Intervention Arm (7-Day Course): Participants will receive 3 mg/kg/day of oral prednisolone for 7 days.
   * Comparator Arm (14-Day Course): Participants will receive 3 mg/kg/day of oral prednisolone for 14 days.
   * In both arms, after 48 hours of in-hospital treatment, participants will be monitored for side effects, and parents will be educated on medication administration and spasm monitoring.
3. Adverse Event Monitoring: Adverse events will be tracked throughout the trial, with particular attention to common side effects associated with prednisolone use, including irritability, weight gain, and gastric irritation. Serious adverse events will be carefully documented and managed.
4. Follow-Up: Follow-up visits will be conducted at 7 days, 14 days, 28 days, 42 days, 3 months, 6 months, and 12 months to monitor spasm control, relapse, and developmental progress. At 24 months, a comprehensive developmental assessment will be conducted to evaluate the long-term effects of the treatment.

Inclusion and Exclusion Criteria:

* Inclusion Criteria: Infants diagnosed with IESS, aged 2 to 24 months, with confirmed spasms either due to a known or unknown aetiology.
* Exclusion Criteria: Infants with a history of other significant neurological conditions, or who are contraindicated for oral prednisolone, including those with uncontrolled systemic infections, significant cardiovascular disease, or severe hypertension.

Data Collection:

Baseline Data: Clinical history, imaging (CT or MRI), and EEG results will be collected to help categorize participants into known or undetermined aetiology groups. A metabolic screening will be conducted for infants with undetermined aetiology.

ELIGIBILITY:
Inclusion Criteria:

* Infants between ages of 3 to 24 months
* Newly confirmed diagnosis of infantile epileptic spasms syndrome made by the referring paediatrician/ paediatric neurologist based on the diagnostic criteria outlined in the recent ILAE classification and definition of epilepsy syndrome with onset in neonates and infants in 2022
* Hypsarrhythmia recorded on pre-treatment EEG. This will be those who show a BASED score of 4 or 5 in a standard EEG

Exclusion Criteria:

* Infants with tuberous sclerosis complex
* Ever treated previously for infantile epileptic spasms syndrome with steroids or other anticonvulsants
* Infants already on steroids or ACTH for any other illness
* Contraindication for the use of high dose steroids such as underlying infection, immune deficiency, hypertension etc.
* Children in critical conditions such as severe infections, congenital heart disease or requiring ventilation or care in an ICU
* Not accompanied by parent/s or parent's inability to complete follow up

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroclinical Remission at Day 14 and Day 28 | Assessed at 14 days and 28 days after treatment initiation.
  This primary outcome measure compares the efficacy of the 7-day versus 14-day oral prednisolone regimens. Electroclinical remission is defined as (1) spasm control-no clinically recognizable spasms for a minimum of 24 consecutive hours as recorded by the caregiver-and (2) EEG remission-disappearance of hypsarrhythmia with the BASED score improved to 3 or less on a standardized 30-minute sleep EEG (with 5 minutes of wakefulness).

SECONDARY OUTCOMES:
Long-Term Spasm Control | Assessed at 42 days, 3 months, 6 months, and 12 months post-treatment.
  This measure evaluates sustained spasm control by documenting the absence of any visible spasms (as observed by caregivers) for at least 72 hours on the day of assessment. It is used to compare the durability of the two treatment regimens over an extended follow-up period.
Spasm Relapse Rate and Time to Relapse | Evaluated continuously over the 12-month follow-up period.
  This outcome captures the relapse rate, defined as the reappearance of clinical spasms in conjunction with the return of hypsarrhythmia on EEG (BASED score of 4 or above), after initial remission. It also records the duration of spasm freedom until the first relapse, providing information on both the frequency and timing of relapse events.
Developmental Outcome at 24 Months | Assessed at 24 months following treatment initiation.
  Neurodevelopmental progress is assessed using the Bayley Scales of Infant and Toddler Development (3rd edition). The measure records deviations from the normative mean (100) across domains (cognition, language, motor skills, social-emotional, and adaptive behavior) and examines correlations with spasm control and relapse status between the treatment arms.
Evolution of Epilepsy | Assessed at 12 months post-treatment.
  This outcome measure tracks the emergence or evolution of other seizure types or epilepsy syndromes beyond infantile spasms. Epilepsy is defined as the occurrence of two or more unprovoked seizures (other than spasms) in a previously spasm-free child. Comparisons between treatment groups will provide insight into long-term seizure evolution.

CONTACTS AND LOCATIONS:
Overall Officials: Jithangi Wanigasinghe, MD, MPhil, Principal Investigator — Department of Paediatrics at the Faculty of Medicine, University of Colombo, Sri Lanka; Carukshi Arambepola, MSc, MD, Principal Investigator — Department of Community Medicine, Faculty of Medicine, University of Colombo, Sri Lanka; Shalini Sri Ranganathan, MD, PhD, Principal Investigator — Department of Pharmacology, Faculty of Medicine, University of Colombo, Sri Lanka; Nimesha Gamhewage, MD, DCH, Principal Investigator — Department of Paediatrics, University of Sri Jayewardenepura, Sri Lanka
Locations (7):
- Sri Lanka (7):
  - Sirimavo Bandaranayake Specialized Children's Hospital, Peradeniya, Central Province
  - Teaching Hospital Anuradhapura, Anuradhapura, North Central Province
  - Teaching Hospital - Jaffna, Jaffna, Northern Province
  - Teaching Hospital - Karapitiya, Galle, Southern Province
  - Lady Ridgeway Hospital for Children, Colombo, Western Province
  - Colombo South Teaching Hospital, Kalubowila, Western Province
  - Colombo North Teaching Hospital, Ragama, Western Province

IPD SHARING:
Plan to Share IPD: No
Since this clinical trial involves infants, who belong to a vulnerable population, strict ethical considerations have been incorporated to ensure data confidentiality and participant protection. All collected data will remain confidential and will be stored securely in a password-protected computer and locked storage, accessible only to the investigators. There is no plan to share individual participant data (IPD).